CLINICAL TRIAL: NCT01271114
Title: Hypertonic Saline and Terlipressin Linked To an Early Goal-Driven Protocol for Septic Shock or Sepsis-Associated Hypotension: A Pilot Trial (HYSATESS)
Brief Title: Hypertonic Saline and Terlipressin for Sepsis-associated Hypotension
Acronym: HYSATESS-p
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Hospital General de Ciudad Real (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Javier Pascual-Ramirez, MD, Hospital General de Ciudad Real
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FISCAM AN-2010/28; 2010-024138-43 (EudraCT Number)
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Septic Shock; Sepsis-associated Hypotension
MeSH Terms: conditions — Shock, Septic | interventions — Saline Solution, Hypertonic; Terlipressin; Saline Solution; Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic Saline and Terlipressin (Experimental)
  Interventions: Drug: Hypertonic Saline and Terlipressin
- Normal Saline and norepinephrine (Active Comparator)
  Interventions: Drug: Normal saline and norepinephrine

INTERVENTIONS:
Drug: Hypertonic Saline and Terlipressin — Hypertonic saline 3% 7mL/Kg (with a maximum 500 mL)triggered by either Systolic Volume Variation or Pulse Pressure Variation more than 10%; Terlipressin infusion (dilution 1mg in 100mL) triggered by MAP below 70 mmHg for a goal MAP above 70 mmHg
  Arms: Hypertonic Saline and Terlipressin
Drug: Normal saline and norepinephrine — Normal saline IV bolus 7mL/kg (with a maximum 500 mL)triggered by either Systolic Volume Variation or Pulse Pressure Variation above 10%; Norepinephrine drip (80 micrograms/mL) to keep MAP at least 70 mmHg
  Arms: Normal Saline and norepinephrine

SUMMARY:
In hypotensive septic patients with controlled source, an hemodynamic management protocol including hypertonic saline (HS)and terlipressin improves MOD (Multiple Organ Dysfunction) Score by at least 3 points compared to the use of physiologic saline and norepinephrine.

The appropriate design for this trial would be factorial. For the time being, will consider de intervention as a whole unit for this pilot study. In the future an appropriately sized factorial multicentric study shall be necessary.

Other goals of the pilot study:

1. HS restores preload parameters adequately
2. HS associated with terlipressin normalizes blood pressure in septic shock
3. HS associated with terlipressin maintains plasma sodium levels 130-155mEq/L
4. There is an inverse relationship between plasma sodium and procalcitonin levels
5. HS increases plasma levels of vasopressin (AVP)
6. HS rises levels of cortisol but not of adrenocorticotropic hormone (ACTH)

ELIGIBILITY:
Inclusion Criteria:

* Criteria of SIRS: at least 2 of 4:

  * Temperature > 38 °c or < 36 ° C
  * More than 90 bpm heart rate
  * Respiratory rate more than 20rpm or PaCO2 less than 32 mm Hg or patient in mechanical ventilation
  * Less than 4000/ mm³ or more than 12000/mm³, or more than 10% leukocyte bands (immature)
* Septic source known demonstrated (or at least of high probability) and controlled (if it is controllable)
* Hematocrit 25% or higher and/or hemoglobin 8 g/dL or higher. If necessary, transfuse RBCs to meet this criteria
* MAP less than 70 mm Hg. Note there is no requirement for adequate preload evidence

Exclusion Criteria:

* Hypernatremia at base-line of 155 mEq/L or greater Hyponatremia at base-line less than 130mEq / L
* Prior endocrine disease affecting to the adrenal-pituitary axis.
* Intracranial Hypertension, brain tumor, seizures, head trauma
* Coronary Artery Disease active over the past year; or evidence of "myocardium at risk" by exercise stress test, pharmacological or positive gammagraphy last year without intervention
* Pregnancy
* Liver disease Child C, End-Stage-Renal-Disease
* Under the age of 18
* Patients with order "do not resuscitate" or with minimal chances to survive

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
MOD (Multiple Organ Dysfunction) Score | daily, as long as the patient stays in the ICU

SECONDARY OUTCOMES:
Hypertonic Saline restores IV fluid response parameters (Pulse Pressure Variation or Systolic Volume Variation) adequately | First 48 hours
Hypertonic Saline associated with terlipressin maintains plasma sodium levels 130-155mEq/L | As long as Hypertonic saline plus terlipressin are in use and one week later
There is an inverse relationship between plasma sodium and plasma procalcitonin levels measured by a negative Pearson coefficient | As long as the patient stays in the ICU
Hypertonic Saline associated with terlipressin normalizes blood pressure in septic shock | First 48 hours
Hypertonic Saline boluses increases plasma levels of vasopressin (AVP) | First week in ICU
Hypertonic Saline use rises levels of cortisol but not of adrenocorticotropic hormone (ACTH) | First week in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pascual Ramírez, Principal Investigator — HGCR; Luis COLLAR VIÑUELAS, MD, Study Chair — HGCR
Locations (1):
- Hospital General de Ciudad Real, Ciudad Real, Ciudad Real, Spain